CLINICAL TRIAL: NCT02409706
Title: Micronutrient Deficiencies in Children and Infants With Congenital Heart Diseases (CHD) Admitted for Cardiac Surgery: A Proof-of-concept Study
Brief Title: Micronutrients in Children in Critical Care With Cardiac Conditions
Acronym: MC5
Status: Completed | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Other Study IDs: GN14KH356; GN14KH356 (Other: NHS Greater Glasgow and Clyde)
Record Dates: First submitted 2015-03-27; First posted 2015-04-07 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Heart Defects, Congenital
Keywords: Paediatric; Critical care; Micronutrients
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood Plasma Red blood cells
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to explore the frequency and types of micronutrient deficiencies in a sample of UK children with CHD using standard and novel markers in blood. The study will also explore whether micronutrient deficiencies increase the risk of complications after heart surgery. This study will identify any nutrient deficiencies that need monitoring in clinical practice.

DETAILED DESCRIPTION:
Congenital heart disease (CHD) is one of the most common birth defects in the UK. Children with CHD are at risk of underfeeding and undernutrition. This is due to both the increased nutritional requirements of the disease and sometimes clinical management, which often hinders delivery of optimal nutrition.There are as yet no studies assessing micronutrient body stores in children with CHD or whether micronutrient deficiencies predict poor clinical outcomes, such as post-operative complications, after major cardiac operations.

This study aims to explore the frequency, types and associations of micronutrient deficiencies in children with CHD using standard and novel markers in blood. The study will also explore whether micronutrient deficiencies increase the risk of complications after heart surgery. This study will identify any nutrient deficiencies that need monitoring in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Infant or child admitted for elective congenital cardiac surgery at the Royal Hospital for Sick Children, Glasgow.
* Aged less than 5 years old

Exclusion Criteria:

* Infant or child admitted for emergency cardiac surgery
* Infant or child whose carer with parental responsibility is unable to communicate in English

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with congenital heart defects who are admitted for elective cardiac surgery at the Royal Hospital for Sick Children, Glasgow.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-08; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Micronutrient Status | Pre- and post- operative: 24-48 hours
  Micronutrient concentrations in plasma and erythrocytes

SECONDARY OUTCOMES:
Postoperative LOS | 1 year
  Length of hospital stay
Postoperative Infectious complications | 1 year
  Incidence of infections
Postoperative ventilator time | 1 year
  Duration of ventilation
Postoperative LICU | 1 year
  Length of stay in PICU

CONTACTS AND LOCATIONS:
Overall Officials: Neil Spenceley, MBChB, Principal Investigator — Royal Hospital for Sick Children, Glasgow
Locations (1):
- Royal Hospital for Sick Children, Glasgow, Glasgow City, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dolk H, Loane M, Garne E. The prevalence of congenital anomalies in Europe. Adv Exp Med Biol. 2010;686:349-64. doi: 10.1007/978-90-481-9485-8_20. PMID 20824455
- [Background] van der Bom T, Zomer AC, Zwinderman AH, Meijboom FJ, Bouma BJ, Mulder BJ. The changing epidemiology of congenital heart disease. Nat Rev Cardiol. 2011 Jan;8(1):50-60. doi: 10.1038/nrcardio.2010.166. Epub 2010 Nov 2. PMID 21045784
- [Background] Nydegger A, Walsh A, Penny DJ, Henning R, Bines JE. Changes in resting energy expenditure in children with congenital heart disease. Eur J Clin Nutr. 2009 Mar;63(3):392-7. doi: 10.1038/sj.ejcn.1602956. Epub 2007 Nov 14. PMID 18000517
- [Background] Mitchell IM, Logan RW, Pollock JC, Jamieson MP. Nutritional status of children with congenital heart disease. Br Heart J. 1995 Mar;73(3):277-83. doi: 10.1136/hrt.73.3.277. PMID 7727190
- [Background] Kogon BE, Ramaswamy V, Todd K, Plattner C, Kirshbom PM, Kanter KR, Simsic J. Feeding difficulty in newborns following congenital heart surgery. Congenit Heart Dis. 2007 Sep-Oct;2(5):332-7. doi: 10.1111/j.1747-0803.2007.00121.x. PMID 18377449
- [Background] Hulst JM, Joosten KF, Tibboel D, van Goudoever JB. Causes and consequences of inadequate substrate supply to pediatric ICU patients. Curr Opin Clin Nutr Metab Care. 2006 May;9(3):297-303. doi: 10.1097/01.mco.0000222115.91783.71. PMID 16607132
- [Background] Bird J, Gentles E, Diamantidi K, Spenceley N, Gerasimidis K. Nutritional intake in a cardiac PICU improved following the introduction of enteral nutrition guidelines. Journal of American Dietetic Association 2013
- [Background] Bird J, Gentles E, Diamantidi K, Alfheeaid H, MacLeod I, Ellis D, Spenceley N, Davidson M, Gerasimidis K. Micronutrient intake in a mixed speciality paediatric intensive care unit. World Congress of Paediatric Intensive Care 2011
- [Background] Gentles E, Bird J, Davidson M, Spenceley N, Ellis D and Macleod I. The impact of fasting, fluid restriction and slow initiation and advancement of enteral feeds on daily energy intake in PICU. Paediatric Intenstive Care Society Annual Conference 2010
- [Background] Briassoulis G, Zavras N, Hatzis T. Malnutrition, nutritional indices, and early enteral feeding in critically ill children. Nutrition. 2001 Jul-Aug;17(7-8):548-57. doi: 10.1016/s0899-9007(01)00578-0. PMID 11448572
- [Background] Vaidyanathan B, Radhakrishnan R, Sarala DA, Sundaram KR, Kumar RK. What determines nutritional recovery in malnourished children after correction of congenital heart defects? Pediatrics. 2009 Aug;124(2):e294-9. doi: 10.1542/peds.2009-0141. Epub 2009 Jul 5. PMID 19581268
- [Background] Padley JR, Cole AD, Pye VE, Chard RB, Nicholson IA, Jacobe S, Baines D, Badawi N, Walker K, Scarfe G, Leclair K, Sholler GF, Winlaw DS. Five-year analysis of operative mortality and neonatal outcomes in congenital heart disease. Heart Lung Circ. 2011 Jul;20(7):460-7. doi: 10.1016/j.hlc.2011.03.009. Epub 2011 Apr 21. PMID 21514216
- [Background] Thiagarajan RR, Laussen PC. Mortality as an outcome measure following cardiac surgery for congenital heart disease in the current era. Paediatr Anaesth. 2011 May;21(5):604-8. doi: 10.1111/j.1460-9592.2011.03580.x. PMID 21481081
- [Background] Cander B, Dundar ZD, Gul M, Girisgin S. Prognostic value of serum zinc levels in critically ill patients. J Crit Care. 2011 Feb;26(1):42-6. doi: 10.1016/j.jcrc.2010.06.002. Epub 2010 Jul 23. PMID 20655701
- [Background] Stoppe C, Schalte G, Rossaint R, Coburn M, Graf B, Spillner J, Marx G, Rex S. The intraoperative decrease of selenium is associated with the postoperative development of multiorgan dysfunction in cardiac surgical patients. Crit Care Med. 2011 Aug;39(8):1879-85. doi: 10.1097/CCM.0b013e3182190d48. PMID 21460705
- [Background] Manzanares W, Biestro A, Torre MH, Galusso F, Facchin G, Hardy G. High-dose selenium reduces ventilator-associated pneumonia and illness severity in critically ill patients with systemic inflammation. Intensive Care Med. 2011 Jul;37(7):1120-7. doi: 10.1007/s00134-011-2212-6. Epub 2011 Mar 29. PMID 21445641
- [Background] Gray A, McMillan DC, Wilson C, Williamson C, O'Reilly DS, Talwar D. The relationship between plasma and red cell concentrations of vitamins thiamine diphosphate, flavin adenine dinucleotide and pyridoxal 5-phosphate following elective knee arthroplasty. Clin Nutr. 2004 Oct;23(5):1080-3. doi: 10.1016/j.clnu.2004.01.013. PMID 15380899
- [Background] Gray A, McMillan DC, Wilson C, Williamson C, O'Reilly DS, Talwar D. The relationship between the acute changes in the systemic inflammatory response, lipid soluble antioxidant vitamins and lipid peroxidation following elective knee arthroplasty. Clin Nutr. 2005 Oct;24(5):746-50. doi: 10.1016/j.clnu.2005.02.008. Epub 2005 Apr 8. PMID 16182038
- [Background] Quasim T, McMillan DC, Talwar D, Vasilaki A, St J O'Reilly D, Kinsella J. The relationship between plasma and red cell B-vitamin concentrations in critically-ill patients. Clin Nutr. 2005 Dec;24(6):956-60. doi: 10.1016/j.clnu.2005.06.004. Epub 2005 Jul 28. PMID 16054730
- [Background] Vasilaki AT, McMillan DC, Kinsella J, Duncan A, O'Reilly DS, Talwar D. Relation between pyridoxal and pyridoxal phosphate concentrations in plasma, red cells, and white cells in patients with critical illness. Am J Clin Nutr. 2008 Jul;88(1):140-6. doi: 10.1093/ajcn/88.1.140. PMID 18614734
- [Background] Vasilaki AT, Leivaditi D, Talwar D, Kinsella J, Duncan A, O'Reilly DS, McMillan DC. Assessment of vitamin E status in patients with systemic inflammatory response syndrome: plasma, plasma corrected for lipids or red blood cell measurements? Clin Chim Acta. 2009 Nov;409(1-2):41-5. doi: 10.1016/j.cca.2009.08.008. Epub 2009 Aug 19. PMID 19698706
- [Background] Vasilaki AT, McMillan DC, Kinsella J, Duncan A, O'Reilly DS, Talwar D. Relation between riboflavin, flavin mononucleotide and flavin adenine dinucleotide concentrations in plasma and red cells in patients with critical illness. Clin Chim Acta. 2010 Nov 11;411(21-22):1750-5. doi: 10.1016/j.cca.2010.07.024. Epub 2010 Jul 24. PMID 20667447
- [Background] Reid D, Toole BJ, Knox S, Talwar D, Harten J, O'Reilly DS, Blackwell S, Kinsella J, McMillan DC, Wallace AM. The relation between acute changes in the systemic inflammatory response and plasma 25-hydroxyvitamin D concentrations after elective knee arthroplasty. Am J Clin Nutr. 2011 May;93(5):1006-11. doi: 10.3945/ajcn.110.008490. Epub 2011 Mar 16. PMID 21411617
- [Background] Talwar D, Quasim T, McMillan DC, Kinsella J, Williamson C, O'Reilly DS. Pyridoxal phosphate decreases in plasma but not erythrocytes during systemic inflammatory response. Clin Chem. 2003 Mar;49(3):515-8. doi: 10.1373/49.3.515. No abstract available. PMID 12600973
- [Background] Gerasimidis K, Talwar D, Duncan A, Moyes P, Buchanan E, Hassan K, O'Reilly D, McGrogan P, Edwards CA. Impact of exclusive enteral nutrition on body composition and circulating micronutrients in plasma and erythrocytes of children with active Crohn's disease. Inflamm Bowel Dis. 2012 Sep;18(9):1672-81. doi: 10.1002/ibd.21916. Epub 2011 Nov 8. PMID 22069243
- [Background] Duncan A, Dean P, Simm M, O'Reilly DS, Kinsella J. Zinc supplementation in intensive care: results of a UK survey. J Crit Care. 2012 Feb;27(1):102.e1-6. doi: 10.1016/j.jcrc.2011.07.083. Epub 2011 Sep 29. PMID 21958977
- [Background] Gerasimidis K, Edwards C, Stefanowicz F, Galloway P, McGrogan P, Duncan A, Talwar D. Micronutrient status in children with IBD: true deficiencies or epiphenomenon of the systemic inflammatory response. J Pediatr Gastroenterol Nutr. 2013 Jun;56(6):e50-1. doi: 10.1097/MPG.0b013e31828f1e86. No abstract available. PMID 23708640
- [Background] Oakes EJ, Lyon TD, Duncan A, Gray A, Talwar D, O'Reilly DS. Acute inflammatory response does not affect erythrocyte concentrations of copper, zinc and selenium. Clin Nutr. 2008 Feb;27(1):115-20. doi: 10.1016/j.clnu.2007.10.003. Epub 2007 Nov 26. PMID 18037540
- [Background] Duncan A, Talwar D, McMillan DC, Stefanowicz F, O'Reilly DS. Quantitative data on the magnitude of the systemic inflammatory response and its effect on micronutrient status based on plasma measurements. Am J Clin Nutr. 2012 Jan;95(1):64-71. doi: 10.3945/ajcn.111.023812. Epub 2011 Dec 7. PMID 22158726
- [Background] Gerasimidis K, Keane O, Macleod I, Flynn DM, Wright CM. A four-stage evaluation of the Paediatric Yorkhill Malnutrition Score in a tertiary paediatric hospital and a district general hospital. Br J Nutr. 2010 Sep;104(5):751-6. doi: 10.1017/S0007114510001121. Epub 2010 Apr 19. PMID 20398432
- [Background] Gerasimidis K, Macleod I, Finlayson L, McGuckin C, Wright C, Flynn D, McGrogan P, Maclean A, Love E, Swinbank I, Mohammed T, McAuley M. Introduction of Paediatric Yorkhill Malnutrition Score--challenges and impact on nursing practice. J Clin Nurs. 2012 Dec;21(23-24):3583-6. doi: 10.1111/j.1365-2702.2012.04164.x. No abstract available. PMID 23145520
- [Background] Stefanowicz FA, Talwar D, O'Reilly DS, Dickinson N, Atkinson J, Hursthouse AS, Rankin J, Duncan A. Erythrocyte selenium concentration as a marker of selenium status. Clin Nutr. 2013 Oct;32(5):837-42. doi: 10.1016/j.clnu.2013.01.005. Epub 2013 Jan 16. PMID 23391458